CLINICAL TRIAL: NCT06636825
Title: Influence of Caffeine on Psychomotor Vigilance and Carbon Dioxide Tolerance During Graded Hypercapnia
Acronym: C3F
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 23-05
Record Dates: First submitted 2024-10-04; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Hypercapnia
Keywords: Caffeine; Carbon dioxide; Cognitive Function
MeSH Terms: conditions — Hypercapnia | interventions — Caffeine

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled crossover trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo (microcrystalline cellulose) capsule taken in a single dose 1 hour prior to graded hypercapnia
  Interventions: Other: Graded hypercapnia; Drug: Placebo
- Experimental (Experimental): 400 mg caffeine capsule taken in a single dose 1 hour prior to graded hypercapnia
  Interventions: Other: Graded hypercapnia; Drug: Caffeine

INTERVENTIONS:
Other: Graded hypercapnia — Volunteers breathe 0%, 2%, 4%, 6%, and 8% CO2 (with 21% O2, balance nitrogen) for 12 minutes each
Drug: Caffeine — 400 mg caffeine capsule taken in a single dose 1 hour prior to graded hypercapnia
  Arms: Experimental
Drug: Placebo — Placebo (microcrystalline cellulose) capsule taken in a single dose 1 hour prior to graded hypercapnia
  Arms: Placebo

SUMMARY:
The aim of this randomized, double-blind, placebo-controlled crossover trial is to determine the effects of caffeine vs. placebo on psychomotor vigilance and carbon dioxide tolerance during graded hypercapnia.

DETAILED DESCRIPTION:
Healthy and fit young adults (men and women) will participate in this study. Participants will perform two primary experimental trials on separate days, one after consuming 400 mg caffeine, and the other after consuming a non-caffeinated placebo. During each trial, participants will breathe increasing levels of inspired CO2 in a stepwise manner (0%, 2%, 4%, 6%, 8% CO2; all with 21% oxygen) during successive 12-minute stages. The endpoints of the graded hypercapnia protocol will be completion of the 8% CO2 stage, voluntary subject termination due to discomfort, or end-tidal CO2 greater than 70 mmHg. The investigators hypothesize that, compared to placebo, caffeine will lower end tidal and arterialized PCO2 and mitigate CO2-mediated decrements in psychomotor vigilance.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18-45
* Body mass index 18.5-30.0 kg m-2
* Body mass 50-100 kg
* In good health as determined by the Office of Medical Support & Oversight (OMSO) General Medical Clearance
* Perform exercise at least 2 times per week
* Willing to abstain from exercise and alcoholic beverages for 24 hours before each study visit.
* Willing to abstain from caffeine for 12 hours prior to all study visits
* Willing to abstain from caffeine for 12 hours after visits 3 and 4
* Willing to remain fasted (no food or fluid other than water) from lights out until after arrival at the laboratory the following morning on each study day (~10 hours)
* Have supervisor approval if permanent party military or a federal employee at U.S. Army Natick Soldier System Center

Exclusion Criteria:

* Females who are pregnant or planning to become pregnant during the study
* Females who are surgically sterile
* History of severe adverse reaction to caffeine (e.g., headache, dizziness, diarrhea, insomnia)
* Taking dietary supplements, prescriptions, or over the counter medication, other than a contraceptive (unless approved by OMSO & PI)
* Abnormal blood count (For example: hemoglobin (Hb) outside of the typical normal values reported by LabCorp in accordance with OMSO (Normal [Hb] Males = 12.6-17.7 g/dL; Females = 11.1-15.9 g/dL) or hematocrit (Hct) outside of the normal ranges (Normal Hct Males = 37.5-51.0%; Females = 34.0-46.6%) levels, presence of abnormal blood chemicals (hemoglobin S or sickle cell traits)
* Any history of pulmonary or cardiovascular disease
* Current diagnosis of asthma (childhood asthma with no recurrence in the last 5 years ok)
* Smokers or nicotine users (unless have quit >1 month prior)
* Current or recent respiratory tract or sinus infections (< 1 month prior)
* Current diagnosis of migraine or recurrent headaches (previous diagnosis with no recurrence in the last 5 years ok)
* Any history of seizures
* Any history of panic disorder
* Blood donation in the previous 8 weeks
* Positive Covid-19 test within the last month (based on self-report)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2023-11-09 (Actual); Primary Completion 2024-09-17 (Actual); Study Completion 2024-09-17 (Actual)

PRIMARY OUTCOMES:
End-tidal CO2 | 60 minutes
  End-tidal CO2 (mmHg)
PVT Performance | 60 minutes
  Psychomotor vigilance (mean reaction time in s)
Carbon dioxide tolerance | 60 minutes
  Time spent in graded hypercapnia protocol (minutes)

SECONDARY OUTCOMES:
Ventilation | 60 minutes
  Ventilation (L/min)
Respiratory Rate | 60 minutes
  Breaths per minute
Tidal volume | 60 minutes
  Tidal volume (L)
Oxygen Consumption | 60 minutes
  Oxygen consumption (L/min)
Carbon dioxide release | 60 minutes
  Carbon dioxide release (L/min)
Heart Rate | 60 minutes
  Heart Rate (Beats per minute)
Blood Pressure | 60 minutes
  Blood pressure (mmHg)
Total Mood Disturbance | 60 minutes
  Profile of Mood States (AU); higher number is worse mood
Arterialized capillary pH | 60 minutes
  pH (unitless)
Arterialized capillary PCO2 | 60 minutes
  Partial pressure of carbon dioxide (mmHg)
Arterialized capillary bicarbonate | 60 minutes
  Bicarbonate (mmol/L))
Dyspnea | 60 minutes
  Borg 0-10 Scale (higher number is more dyspnea)
Discomfort | 60 minutes
  Borg 0-10 Scale (higher number is more discomfort)
Headache | 60 minutes
  100mm visual analog scale (higher number is worse headache)
Plasma caffeine | 60 minutes
  Plasma caffeine (ug/mL)
Plasma theobromine | 60 minutes
  Plasma theobromine (ug/mL)
Plasma theophylline | 60 minutes
  Plasma theophylline (ug/mL)
Plasma paraxanthine | 60 minutes
  Plasma paraxanthine (ug/mL)

CONTACTS AND LOCATIONS:
Locations (1):
- US Army Research Institute of Environmental Medicine, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-02-26): https://cdn.clinicaltrials.gov/large-docs/25/NCT06636825/ICF_000.pdf